CLINICAL TRIAL: NCT03311204
Title: The Effect and Duration of Efficacy of Eyelid Margin Debridement on Signs and Secretions of Eyelids, Tear Film and Discomfort in Contact Lens Wearers
Brief Title: The Effect of Eyelid Margin Debridement on Contact Lens Discomfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Jaya Sowjanya Siddireddy, Ms, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UNewSouthwales
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Contact Lens Discomfort
Keywords: Eyelid margin; Tear Film; Debridement; Contact Lens; Ocular Discomfort

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, cross-over, open-label interventional study
Who Masked: Outcomes Assessor
Masking Description: The clinical signs are photographed and an outcomes accessor grades the clinical signs. This process ensures that there is no bias in recording the results. This method was specially chosen, due to the lack or inability to mask the treatment procedures, due to their nature of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microblepharon Exfoliation (Experimental): This treatment is provided using BlephEx tool from Optimed Pty Ltd.
  Interventions: Device: BlephEx
- Eyelid cleansing using Lid Hygenix (Experimental): Foam-based hypoallergenic cleanser used as a control treatment in this study.
  Interventions: Other: Lid Hygenix

INTERVENTIONS:
Device: BlephEx — BlephEx is an instrument that contains a hand piece used to spin a medical grade micro-sponge along the edge of eyelids and lashes that helps in removing scurf and debris from eyelids and helps in exfoliating the lids. A new micro-sponge will be used for every subject to avoid cross-contamination. This procedure lasts for 6-8 mins.
  Arms: Microblepharon Exfoliation
Other: Lid Hygenix — Foam-based hypoallergenic cleanser used to clean eyelid margins is used as a control intervention for the study.
  Arms: Eyelid cleansing using Lid Hygenix

SUMMARY:
In this study, clinical variables related to eyelids that potentially have an effect on contact lens discomfort will be investigated such as eyelid signs and secretions, eyelid sensitivity, eyelid microbiome, Demodex infestation and tear film properties. The main aim of this study is to understand the duration of efficacy of debridement of the eyelid margin and its impact on various eyelid signs (such as lid wiper epitheliopathy, lid-parallel conjunctival folds, eyelid sensitivity, meibomian gland morphology and meibum secretions, palpebral conjunctival reaction, eyelid microbiome and Demodex infestation, tear properties (both biophysical properties such as tear volume, tear meniscus height, tear evaporation, tear osmolarity and tear breakup time; and biochemical properties that are tear lipid analysis). To observe these variables, this study employs a cross-sectional design to study the effect of treatment at three instances, that is at baseline and two follow-up visits.

DETAILED DESCRIPTION:
Contact lens discomfort (CLD) is a substantial problem experienced frequently by contact lens wearers and it is the primary factor associated with permanent discontinuation of lens wear. Studies report that between 43% and 72% of contact lens wearer's dropout due to discomfort. Reducing the number of contact lens (CL) patient dropouts has been a continuing challenge for eye care professionals. With more than 125 million contact lens wearers around the world, patient discontinuations can have a considerable economic impact on an eye care practice.

Definition: Contact lens discomfort is a condition characterized by episodic or persistent adverse ocular sensations related to lens wear, either with or without visual disturbance, resulting from reduced compatibility between the contact lens and the ocular environment, which can lead to decreased wearing time and discontinuation of contact lens wear.

Inferences from our earlier study (HC15119) showed that eyelid margin debridement significantly improves eyelid signs, tear film properties and comfort in contact lens wearers. But the previous study did not consider the duration of efficacy as the subjects were only followed up once after 7-10days from treatment. Observing subjects more frequently will help us understand the duration of efficacy of debridement therapy. Also, the previous study did not examine the biochemical changes to tear film lipids that are produced by the eyelids.

It is hypothesized that debridement of eyelid margins improves lipid secretions that then help to form a stable lipid layer over ocular surface, thereby improving the tear evaporation dynamics and comfort in contact lens wearers.

Aim: The aim of the study is to observe the duration of efficacy of debridement of the eyelid margins in improving secretions from eyelid glands and whether the debridement helps to form a stable tear film over ocular surface, thereby improving comfort in contact lens wearers.

Objectives: To determine the effect of BlephEx - debridement therapy (an in-office eyelid treatment) on eyelid signs and secretions, tear film and contact lens discomfort.

To observe differences in discomfort in contact lens wearers To determine the duration of efficacy of BlephEx debridement therapy in contact lens wearers, by following up after 12-15 days and 22-25days from the baseline (Treatment) visit.

Methods: The study employs cross-sectional study design, to observe the effect of treatment at three instances, one baseline (treatment) visit and two follow-up visits. At the baseline visit, informed consent will be obtained from the subjects and assessment of the study variables will be performed. Participants will undergo treatment on the same day with BlephEx. At baseline, the measurements are performed prior to treatment to record preliminary scores and then treatment is performed. Participants are asked to return to the clinic for follow-up visits during which no treatment will be performed, but variables are assessed to determine the difference from baseline measurements. The 2nd visit will be after 12 -16 days after the baseline visit. The last follow-up will be 22-26 days after the baseline visit. All study variables will be assessed during all three visits to the clinic.

Treatment Procedure: BlephEx is an instrument that contains a handpiece used to spin a medical grade micro-sponge along the edge of eyelids and lashes that helps in removing scurf and debris from eyelids and helps in exfoliating the lids. A new micro-sponge will be used for every subject to avoid cross-contamination. This procedure lasts for 6-8 mins.

Lid Hygenix is a commercially available formulated hypoallergenic foam cleanser will be used to moisten the BlephEx debridement tips.

Both the products are commercially available. The procedure is safe, painless and regularly performed by optometrists.

'Participant information sheet and informed consent' and 'web-based survey for the end of the day discomfort rating' will be sent out in the form of an email. Participants who are interested in participation will respond to the survey and results will be used only after the subject signs the informed consent in the presence of the investigator, during the baseline visit. This survey response will be used as baseline data for the end of the day discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or above
* Understand their rights as a research subject
* Willing and able to sign a statement of informed consent
* Normal ocular status, defined as a minimum of 20/40 visual acuity in each eye; clear corneas without scarring, opacities, or vascularization, as determined by biomicroscopic examination
* Normal external examination
* Normal puncta without punctal plugs
* Ability to cooperate with the required procedures of diagnostic agent installation, eyelid eversion, and examination.
* Contact lens wearers who have worn lenses for at least 6 months, used contact lenses for 3 weeks before the evaluation visit and used these lenses at least four times a week. These contact lens wearers will be on daily wearing modality, where the subject is supposed to wear it for at least for 6 hours, only during the day and remove the lenses during sleep.

Exclusion Criteria:

* Any ocular or systemic disease that might influence the tear film and especially subjects with a history of episodes of epilepsy.
* Subjects with eyelid inflammation of more than grade 2 will be excluded from the study as they need therapeutic intervention.
* All conjunctival abnormalities, including pingueculae greater than 1 mm in diameter, location closer than 2 mm to the limbus, or elevated more than 0.2 mm
* All forms of conjunctivitis, including allergic conjunctivitis
* Fluorescein corneal staining of grade 2 or more, after a single installation of non-preserved fluorescein solution followed by examination 1 minute after installation
* Current ocular infection or treatment of such infections with ocular or systemic medications
* Current use of any prescription or non-prescription ocular or systemic medications, including antihistamines
* Use of artificial tear preparations during the period 2 hours before the examination
* Use of any ocular ointment during the 3 days before the examination
* Any history of ocular surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Lid Wiper Epitheliopathy | 5 minutes
  The eyelids will be examined using a slit lamp before and after instillation of sodium fluorescein. This stain helps to disclose changes to the eyelid surface .

SECONDARY OUTCOMES:
Discomfort Rating - CLDEQ-8 Questionnaire | 5 minutes
  Discomfort will be measured using the CLDEQ-8 questionnaire that involves questions about participants' experience of discomfort. This will be employed on all the study visits in the clinic.
End of the Day Discomfort Rating | 30 minutes
  End of the day discomfort will be assessed using a visual analog scale, where questions will be posed to participants about their level of comfort with contact lens wear at a specific time of day. This questionnaire will be a web-based survey, sent in the form of an email on the day before the baseline visit, and day 4, 9, 14, 19 and 24 from baseline visit.
Tear Analysis | 15 minutes
  Change in tear lipids at day 4, 9, 14, 19 and 24 compared to baseline
Meibum Analysis | 10 minutes
  Change in meibum lipids at day 4, 9, 14, 19 and 24 compared to baseline.
Meibography | 5 minutes
  Meibomian gland (glands in eyelids) morphology will be compared at day 4, 9, 14, 19 and 24 compared to baseline.
Demodex Infestation | 15 minutes
  Highly magnified images of eyelids will be captured with a microscope to count the number of Demodex on eyelids. these images will be compared at day 4, 9, 14, 19 and 24 compared to baseline.
Lid Microbiota | 5 minutes
  Change in colony forming units of cultivable eyelid microbiota will be compared at day 4, 9, 14, 19 and 24 compared to baseline.
LipiView Interferometry | 10 minutes
  The change in absolute thickness of the tear film lipid layer will be compared at day 4, 9, 14, 19 and 24 compared to baseline.
Lid Sensitivity | 5 minutes
  Change in eyelid sensitivity assessed using Cochet Bonnet aesthesiometer will be compared at day 4, 9, 14, 19 and 24 compared to baseline.
Tear Osmolarity | 5 minutes
  Change in tear osmolarity using TearLab osmometer will be compared at day 4, 9, 14, 19 and 24 compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Willcox, D Sc, Study Chair — University of New South Wales
Locations (1):
- University of New South Wales, Kensington, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
All participants will be given a unique study identification code. Data will be de-identified at the time of collection such that only patient initials and a study identification number will be used to identify the data for each patient. Any data included in reports, publications or presented at meetings will be provided in the form of group responses or study identity numbers, such that the participants cannot be identified. Personal and health information (either identifiable or potentially identifiable) about individuals will not be disclosed to any external parties without the individual's consent unless required by law. The unique study identification code can be broken by the research team if required (re-identifiable).